CLINICAL TRIAL: NCT00032227
Title: Carpal Tunnel Syndrome: Diagnosis and Treatment Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Jeffrey G. Jarvik, MD, MPH, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P60AR048093 (NIH); P60AR048093 (NIH); NIAMS-075
Record Dates: First submitted 2002-03-12; First posted 2002-03-13 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Release; MR Nerve Imaging; Wrist MRI
MeSH Terms: conditions — Carpal Tunnel Syndrome

ARMS (2):
- 1 (Experimental): Surgical release of CTS
  Interventions: Procedure: Early Carpal Tunnel Release for Mild or Moderate CTS; Other: MR Nerve Imaging for CTS
- 2 (Active Comparator): Non-surgical treatment for CTS (splint, physical therapy, ultrasound)
  Interventions: Procedure: Early Carpal Tunnel Release for Mild or Moderate CTS; Other: MR Nerve Imaging for CTS

INTERVENTIONS:
Procedure: Early Carpal Tunnel Release for Mild or Moderate CTS — Either open or endoscopic surgery
Other: MR Nerve Imaging for CTS — New diagnostic test for CTS to directly image the median nerve

SUMMARY:
The Carpal Tunnel Syndrome Diagnosis and Treatment Trial is project #1 of the Multidisciplinary Clinical Research Center focused on upper extremity pain. It is a randomized trial comparing surgical and nonsurgical treatments for patients with early, mild to moderate carpal tunnel syndrome. In addition the study will evaluate the ability of a new magnetic resonance (MR) technique at predicting who will likely benefit from carpal tunnel syndrome (CTS) surgery.

DETAILED DESCRIPTION:
While there is good evidence that patients with severe CTS benefit from surgery, there is less evidence of a benefit for patients with mild to moderate disease. However, mild to moderate disease still accounts for important disability. Electrodiagnostic studies (EDS) have not been shown to accurately predict outcomes for patients with CTS. Recent advances in MR permit high-resolution neurographic imaging of the median nerve, and pilot data suggest that wrist MRI might be a better predictor of outcome than EDS. Thus, wrist MRI has the potential for playing a major role in the treatment of patients with CTS. We will test two main hypotheses: 1) that select patients with early, mild or moderate CTS benefit more from early surgery than with conservative therapy; and, 2) that wrist MRI accurately identifies those patients more likely to benefit from surgery. We will perform a randomized, controlled treatment trial nested within a prospective cohort as our study design.

ELIGIBILITY:
Inclusion Criteria:

* Paresthesias involving 2 digits on hand diagram
* Willingness and ability to complete interviews

Exclusion Criteria:

* Evidence of denervation on EDS
* Abnormal 2-pt discrimination or thenar atrophy
* Prior wrist surgery or acute external trauma
* MRI contraindications
* Metallic hardware in wrists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2002-08; Primary Completion 2007-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Carpal Tunnel Syndrome Assessment Questionnaire- function scale | 12 months

SECONDARY OUTCOMES:
CTSAQ symptom scale | 12 months
CTSAQ-function | 3 months
CTSAQ-symptom | 3 months
SF36 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey G. Jarvik, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Jarvik JG, Yuen E. Diagnosis of carpal tunnel syndrome: electrodiagnostic and magnetic resonance imaging evaluation. Neurosurg Clin N Am. 2001 Apr;12(2):241-53. PMID 11525204
- [Background] Grant GA, Britz GW, Goodkin R, Jarvik JG, Maravilla K, Kliot M. The utility of magnetic resonance imaging in evaluating peripheral nerve disorders. Muscle Nerve. 2002 Mar;25(3):314-31. doi: 10.1002/mus.10013. PMID 11870709
- [Background] Aagaard BD, Lazar DA, Lankerovich L, Andrus K, Hayes CE, Maravilla K, Kliot M. High-resolution magnetic resonance imaging is a noninvasive method of observing injury and recovery in the peripheral nervous system. Neurosurgery. 2003 Jul;53(1):199-203; discussion 203-4. doi: 10.1227/01.neu.0000069534.43067.28. PMID 12823890
- [Background] Jarvik JG, Yuen E, Haynor DR, Bradley CM, Fulton-Kehoe D, Smith-Weller T, Wu R, Kliot M, Kraft G, Wang L, Erlich V, Heagerty PJ, Franklin GM. MR nerve imaging in a prospective cohort of patients with suspected carpal tunnel syndrome. Neurology. 2002 Jun 11;58(11):1597-602. doi: 10.1212/wnl.58.11.1597. PMID 12058085
- [Background] Jarvik JG, Yuen E, Kliot M. Diagnosis of carpal tunnel syndrome: electrodiagnostic and MR imaging evaluation. Neuroimaging Clin N Am. 2004 Feb;14(1):93-102, viii. doi: 10.1016/j.nic.2004.02.002. PMID 15177259
- [Background] Martin BI, Levenson LM, Hollingworth W, Kliot M, Heagerty PJ, Turner JA, Jarvik JG. Randomized clinical trial of surgery versus conservative therapy for carpal tunnel syndrome [ISRCTN84286481]. BMC Musculoskelet Disord. 2005 Jan 18;6:2. doi: 10.1186/1471-2474-6-2. PMID 15656907
- [Background] Storm S, Beaver SK, Giardino N, Kliot M, Franklin GM, Jarvik JG, Chan L. Compliance with electrodiagnostic guidelines for patients undergoing carpal tunnel release. Arch Phys Med Rehabil. 2005 Jan;86(1):8-11; quiz 180. doi: 10.1016/j.apmr.2004.02.027. PMID 15640981
- [Derived] Jarvik JG, Comstock BA, Kliot M, Turner JA, Chan L, Heagerty PJ, Hollingworth W, Kerrigan CL, Deyo RA. Surgery versus non-surgical therapy for carpal tunnel syndrome: a randomised parallel-group trial. Lancet. 2009 Sep 26;374(9695):1074-81. doi: 10.1016/S0140-6736(09)61517-8. PMID 19782873